CLINICAL TRIAL: NCT03429582
Title: Comparison of Cervical Intraepithelial Neoplasia 2/3 Treatment Outcomes With a Portable LMIC-adapted Thermal Ablation Device vs. Gas-based Cryotherapy
Brief Title: Comparison of Cervical CIN II/III Treatment Outcomes With Thermal Ablation Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Basic Health International (Other); WISAP Medical Technologies GMBH (Unknown); University of Southern California (Other); Medical College of Wisconsin (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-1385; 1R01CA218195-01A1 (NIH)
Record Dates: First submitted 2018-01-25; First posted 2018-02-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Human Papilloma Virus; Thermoablation; Thermocoagulation; Cryotherapy; Cervica Pre-cancer; Low and Middle Income Countries (LMICs)
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard C02 Cryotherapy (Active Comparator): Standard therapy using carbon dioxide for freezing of tissue
  Interventions: Device: Standard C02 Cryotherapy
- Single Tip Thermoablation (Experimental): Thermoablator outfitted with a 19mm conical tip
  Interventions: Device: Single Tip Thermoablation
- Multiple Tip Thermoablation (Experimental): Thermoablator outfitted with detachable probes
  Interventions: Device: Multiple Tip Thermoablation

INTERVENTIONS:
Device: Standard C02 Cryotherapy — Standard therapy using carbon dioxide for freezing of tissue
  Arms: Standard C02 Cryotherapy
Device: Single Tip Thermoablation — Thermoablator outfitted with a 19mm conical tip
  Arms: Single Tip Thermoablation
Device: Multiple Tip Thermoablation — Thermoablator outfitted with detachable probes
  Arms: Multiple Tip Thermoablation

SUMMARY:
The purpose of this academic-industrial partnership will be to compare two thermoablation modalities using devices adapted to low and middle income countries (LMICs) to traditional CO2-based cryotherapy for the treatment of cervical precancer. The investigators will investigate whether the cure rates of cervical intraepithelial neoplasia 2 and more severe diagnoses (CIN2+) with these devices are non-inferior compared to that of conventional cryotherapy. The results of this study will affect other research areas by serving as a springboard to exploring treatment alternatives that are amenable to low-resource settings and thus will reach the most vulnerable populations.

DETAILED DESCRIPTION:
The standard treatment for cervical pre-cancer is gas-based cryotherapy, the freezing of tissue to ablate (destroy) lesions. Although cryotherapy is relatively simple to perform, the necessary gas tanks are generally expensive, difficult to obtain and transport, and pose a danger of explosion. An urgent need exists for a point-of-care treatment technology that is accessible, portable, and inexpensive. An alternative ablative procedure in use since the 1970s is thermoablation (also known as cold coagulation or thermocoagulation), which utilizes heat to destroy pre-cancer. Despite its long-standing use, there are no standardized guidelines for thermoablation. There is also little data on patient and provider acceptability, potential side effects, and the impact of different treatment protocols on quality of life. For these reasons, international and national agencies have been hesitant to adopt the technique as an alternative to cryotherapy. The purpose of this research study is to develop a patient-centered thermoablation protocol that is simple, safe, and effective.

Currently, the most common treatment technique for thermoablation involves a multiple-tip protocol, which uses differently shaped probe-tips to cover the affected area. This technique requires a considerable degree of expertise, and may not be the most appropriate strategy for settings where highly trained healthcare providers are scarce. In collaboration with WiSAP Medical Technology (Brunnthal, Germany), the manufacturer of the most widely used thermoablator, the investigators modified the original device to meet the needs of low-resource settings. The LMIC-adapted thermoablator is lightweight, portable, and easy to operate. The investigators will further modify the LMIC-adapted thermoablator to test the non-inferiority of two thermoablation treatment approaches against the standard of care (i.e. gas-based cryotherapy). The experimental approaches include:

1. Single tip: A 19mm conical tip with a nipple is applied to the cervix for 40-seconds at 100ºC, a single application of which should ablate the squamocolumnar junction (SCJ) in the majority of women. In the rare instance that the SCJ is not completely ablated, additional 20 second applications can be applied, or
2. Multiple tips: A narrow nipple shaped tip at 100ºC is placed in the endocervix for 20 seconds. This is followed by the placement of a 12 mm flat tip at 100ºC on the ectocervix for as many 20-second applications as necessary to ablate the entire SCJ.

These will be tested against traditional CO2 cryotherapy treatment using a MedGyn device in a standard double-freeze procedure (3 minute freeze, 5 minute thaw, 3 minute freeze).

Women will be recruited at colposcopy clinics run by the Ministry of Health and the Mexican Institute of Social Security (Instituto Mexicano del Seguro Social) in the Mexico City metropolitan region. Eligible women will be those over the age of 18, who are able and willing to provide informed consent and a reliable or permanent address, and with a biopsy-confirmed CIN2+ diagnosis. Women wo are pregnant, plan to become pregnant during the study duration, with a history of total hysterectomy, past surgeries destructive to the cervix within the last 5 years, with a disfigure or hard-to-reach cervix, and those with contraindications for ablative treatment will be excluded from the study.

The investigators will approach 1,602 women with CIN2+ during a four-year enrollment phase (48 months). Assuming an 80% participation rate, approximately 1,282 women will be enrolled; of these, 1,155 (90%) will be eligible for ablation treatment (i.e. no contraindications) and 129 will be ineligible and undergo alternative treatments (i.e. LEEP or invasive cancer treatment). The investigators estimate that approximately 20% will be lost to follow-up at the 12-month visit, resulting in complete data on a total of 924 women (57.7% of 1,602) treated with CO2-based cryotherapy, single-tip thermoablation, or multiple-tip thermoablation. The investigators will monitor the percentages of ineligible women, contraindications, and loss to follow-up in real time and adjust recruitment accordingly to achieve the target sample size.

The clinical endpoint of the study will be residual disease at the 12-month follow-up visit as determined by colposcopy, four-quadrant biopsy, and endocervical curettage (ECC). HPV testing will also be performed at this visit to differentiate between persistent or new infection. Cytology, VIA and care HPV tests will also be performed to evaluate the most effective post treatment screening strategy.

At a pre-treatment visit, consented women will receive a pregnancy test as part of the eligibility criteria for enrollment in the study. Pre-vaginal cultures will be collected to be analyzed for bacterial vaginosis, yeast, gonorrhea and chlamydia. The same cultures will be collected at a 6-week follow-up visit. Consented women will be enrolled and undergo a pelvic exam and visual inspection of the cervix following placement of diluted acetic acid on the cervix. Images of the cervix will be taken with a mobile colposcopy device will be taken before and after treatment. Women will be asked to evaluate their pain level after speculum insertion, immediately before treatment, and immediately after treatment. These women will also complete a quality of life assessment. Women deemed ineligible for cryotherapy will undergo LEEP immediately. In the case of suspected cancer, women will be appropriately referred.

Six weeks post-treatment, women who return for a visit for evaluation of treatment side effects; these women will be administered a post-treatment patient satisfaction survey, and complete a questionnaire to assess the presence of pain or cramps, bleeding, stenosis, watery discharge, malodorous discharge and be evaluated for evidence of cervicitis. In addition, vaginal cultures will be collected and analyzed for bacterial vaginosis, yeast, gonorrhea, and chlamydia.

One year post-treatment, women will return for a follow-up visit to determine residual disease, which is the primary endpoint. Residual disease will be determined by colposcopy and four-quadrant biopsies. In addition, VIA, cytology, and high-risk HPV DNA testing with careHPV will be performed. Genotyping and next-generation sequencing will be repeated to differentiate between persistent and new infections. The investigators will evaluate sensitivity of VIA, cytology, and HPV testing post-treatment. Women will be asked to again complete the quality of life assessment and treatment acceptability instrument. Women diagnosed with recurrent/untreated CIN2+ on biopsy will be asked to return to undergo LEEP. Women with suspected cancer on biopsy will be referred to the local cancer hospital for standard of care.

ELIGIBILITY:
Criteria for inclusion

* Women aged 18 and older
* Biopsy results of CIN2, CIN2-3, CIN3, or high-grade CIN not otherwise specified
* Willing and able to provide informed consent
* Willing and able to provide permanent or reliable address

Criteria for exclusion

* Pregnant or plans to become pregnant during study
* History of total hysterectomy (verified by medical record or pelvic evaluation)
* Previous surgery destructive to the cervix within the last 5 years
* Patient not eligible for cryotherapy or thermoablation (lesion >75% of cervix, lesion extends into canal or there is suspicion for invasive cancer)
* Cervix shape disfigured or hard to reach

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1154 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Residual CIN2+ diagnosis of recurrent and or untreated cervical intraepithelial neoplasia grade 2 or with cervical cancer diagnosis Diagnosis of recurrent and or untreated cervical intraepithelial neoplasia grade 2 or with cervical cancer diagnosis | 12-months post treatment
  To compare CIN2+ cure rates 12-months post-treatment for CO2-based cryotherapy and both single versus multiple tips thermoablation strategies

SECONDARY OUTCOMES:
Patient's pain assessed using the Wong-Baker FACES scale | Immediately after speculum insertion, immediately before treatment, and immediately after treatment
  Functional Assessment of Chronic Illness Therapy for Patients with Cervical Dysplasia Version 4 (FACIT-CD). Consists of 5-subscales listed below. For all subscales and the scale, 0 is the worst outcome, higher scores are better outcomes. All subscales are summed.
  Subscale ranges are as follows: Physical well-being:0 to 32, Treatment satisfaction:0 to 16, General perceptions:0 to 28, Emotional well-being:0 to 44, Relationship support: 0 to 16 Wong-Baker FACES® Pain Rating Scale, construct being measured is pain for anyone over the age of 3. Scale range: Minimum = 0, Maximum = 10. For each scale range, what is a better or worse outcome: 0 is a better outcome (no pain), higher scores are worse outcomes, and 10 is the worst outcome (worst pain). There are no subscales.

OTHER OUTCOMES:
Patient's satisfaction with treatment assessed with the FACIT-CD questionnaire (FACIT Measurement System) | At enrollment, 6-week visit, and 12-month follow-up visit
  FACIT-CD Version 4: 5-subscales. For all subscales and the scale, 0 is the worst outcome, higher scores are better outcomes. All subscales are summed. Subscale ranges are as follows: Physical well-being:0 to 32, Treatment satisfaction: 0 to 16, General perceptions: 0 to 28, Emotional well-being:0 to 44, Relationship support: 0 to 16
Patient's hope for the future using the Herth Hope Index | At enrollment and at 12-month follow-up visit
  Herth Hope Index. The construct is hope in adults in clinical settings. Scale ranges: 1 to 4. For the total index, 12 is the worst outcome. Higher scores are better outcomes. There are no subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Cremer, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- Peking University Shenzhen Hospital, Shenzhen, China
- Hospital Nacional de la Mujer, San Salvador, El Salvador

IPD SHARING:
Plan to Share IPD: No